CLINICAL TRIAL: NCT00922688
Title: Dipeptide Alanyl Glutamine and Postoperative Insulin Resistance in Colon Carcinoma Patients
Acronym: AIRCo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: H. Cakir, Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AIRCo05.02.2009/2
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-11

CONDITIONS: Colon Carcinoma
Keywords: Dipeptide Alanyl-Glutamine; Insulin sensitivity; Intracellular signaling; Antioxidant/oxidant parameters; Lipolysis; Inflammatory response in the liver
MeSH Terms: conditions — Colonic Neoplasms; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dipeptiven Arm Enteral (Active Comparator)
  Interventions: Drug: Dipeptide Alanyl-Glutamine
- Placebo Arm Enteral and Intravenously (Placebo Comparator)
  Interventions: Drug: Placebo
- Dipeptiven ARM Intravenously (Active Comparator)
  Interventions: Drug: Dipeptide Alanyl-Glutamine

INTERVENTIONS:
Drug: Dipeptide Alanyl-Glutamine — Intravenous supplementation of the dipeptide alanyl-glutamine is started 24 hours prior to surgery (dosage glutamine: 0,5 g/kg/day, and continued 24 hours postoperatively.
  Arms: Dipeptiven ARM Intravenously
Drug: Placebo — Intravenous and enteral supplementation of placebo is started 24 hours prior to surgery and continued 24 hours postoperatively.
  Arms: Placebo Arm Enteral and Intravenously
Drug: Dipeptide Alanyl-Glutamine — Enteral supplementation of the dipeptide alanyl-glutamine is started 24 hours prior to surgery (dosage glutamine: 0,5 g/kg/day, and continued 24 hours postoperatively.
  Arms: Dipeptiven Arm Enteral

SUMMARY:
Rationale: It is well known that insulin resistance occurs after mediocre and intensive surgery, such as colon cancer surgery. Disturbances in insulin action negatively affect the postoperative recovery, either by prolonging the capacity of the body to regain normal function, or by increasing the metabolic stress and the risk for complications. Several studies have shown that focusing therapies on improving insulin resistance is successful. Experimental studies have shown that antioxidant agents, like glutamine (a precursor of glutathione), improve insulin sensitivity. The hypothesis of this study is that perioperative parenteral or enteral administration of glutamine, given as the dipeptide alanyl-glutamine, will reduce or prevent postoperative insulin resistance in colon cancer patients. The study will also be focused on the different routes of administration, because of the expected differential metabolic effects.

Objective: The investigators' primary objective is to study whether intravenous or enteral administration of the dipeptide alanyl-glutamine will reduce or prevent postoperative insulin resistance in colon cancer patients.

Study design: A double-blinded, placebo controlled randomised, pilot study at the Surgery Department of the Medical Center Alkmaar.

Study population: Thirty patients of male gender and any ethnicity, who will undergo elective open abdominal colon surgery for colon cancer, aged 18-75 years.

Intervention: Patients will receive dipeptide alanyl-glutamine intravenously or enterally, starting 24 hours prior to surgery, until 24 hours after surgery in the dosage of 0.5 g/kg/day, or saline (control group), for the same period of time.

Main study parameters/endpoints: The main study parameter is postoperative insulin resistance. Secondary study parameters are lipolysis, oxidative stress and glucoregulatory hormones. Muscle, liver and fat biopsies will be taken to study insulin sensitive as well as inflammatory pathways.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Colon cancer patients scheduled for elective open abdominal surgery
* Capable of giving informed consent

Exclusion Criteria:

* Patients who are participating in another clinical trial
* Unable to receive oral intake
* Major malabsorption disorder of the gut
* Patients with diabetes mellitus
* BMI above 30 kg/m2
* Use of certain medication: thyroid medication, corticosteroids, diuretic medication
* Known bleeding disorders or increased PTT and or APTT
* Any medical condition except for colon cancer

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
The effect of intravenously and enterally administered dipeptide alanyl-glutamine preoperatively on postoperative insulin resistance in colon cancer patients.given, on postoperative insulin resistance in colon cancer patients. | Before and 1 day after surgery

SECONDARY OUTCOMES:
The effect of the dipeptide alanyl-glutamine on components of the insulin signalling cascade in muscle tissue. | Before and 1 day after surgery
The effect of the dipeptide alanyl-glutamine on the systemic inflammatory response as well as on inflammatory pathways in muscle. | Before and 1 day after surgery
The effect of the dipeptide alanyl-glutamine on the amino acid concentration in muscle tissue. | Before and 1 day after surgery
The effect of the dipeptide alanyl-glutamine on antioxidant/oxidant parameters in the circulating compartment. | Before and 1 day after surgery
The effect of dipeptide alanyl-glutamine on the inflammatory response in the liver | During surgery
The effect of dipeptide alanyl-glutamine on lipolysis. | Before and 1 day after surgery
The effect of dipeptide alanyl-glutamine on key enzymes involved in glucose production. | Before and 1 day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander PJ Houdijk, MD,PhD, Study Director — MCA Alkmaar
Locations (1):
- Medical Center Alkmaar, Alkmaar, North Holland, Netherlands